CLINICAL TRIAL: NCT03551093
Title: A Multicenter, Single Arm Trial to Assess Safety and Signal of Efficacy of the Ischemic Stroke System (ISS), as an Adjunct to Standard of Care in Subjects With Mild Acute Ischemic Stroke
Brief Title: THE IMPACT- 24M TRIAL (IMPlant Augmenting Cerebral Blood Flow in Mild Strokes Trial 24 Hours From Stroke Onset)
Acronym: ImpACT-24M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BrainsGate (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP0050613
Record Dates: First submitted 2018-05-17; First posted 2018-06-11 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-04

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; Mild Acute Ischemic Stroke; Safety; Signal of Efficacy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: This will be a multi-center, adjunctive to Standard of Care, single arm study, which includes the following steps:
  1. Screening (day 1)
  2. Implantation (day 1)
  3. Treatment and symptom assessment (days 1-5)
  4. Device Positioning and Removal (day 5)
  5. Discharge/Final Visit (day 7-10)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Population (Experimental): The ISS is intended to deliver electrical stimulation to the nerves within the greater palatine canal and pterygopalatine fossa.
  Interventions: Device: ISS SPG stimulation

INTERVENTIONS:
Device: ISS SPG stimulation — The ISS is intended to deliver electrical stimulation to the nerves within the greater palatine canal and pterygopalatine fossa (SPG).

SUMMARY:
Study Population:

Subjects with Mild Acute Ischemic Stroke in the anterior circulation within 24 hours from onset.

Study objectives:

1. Identify the personal stimulation level for each patient based on physiological biomarkers
2. Identify improvement in stroke symptoms during ISS treatment at the personal stimulation level

DETAILED DESCRIPTION:
A Multicenter, Single Arm Trial to Assess Safety and Signal of Efficacy of the Ischemic Stroke System (ISS), as an Adjunct to Standard of Care in Subjects with Mild Acute Ischemic Stroke

Study Duration:

The expected total duration of the study for each subject is up to 10 days as follows:

Enrollment: up to 24 hours Treatment: Implantation, 5 Days of SPG stimulation and Standard of care Final Visit: 7 days after enrollment

Study Population:

Subjects with Mild Acute Ischemic Stroke in the anterior circulation within 24 hours from onset.

Study Objectives:

1. Identify the personal stimulation level for each patient based on physiological biomarkers
2. Identify improvement in stroke symptoms during ISS treatment at the personal stimulation level

Study Design:

This will be a multi-center, adjunctive to Standard of Care, single arm study, which includes the following steps:

1. Screening (day 1)
2. Implantation (day 1)
3. Treatment and symptom assessment (days 1-5)
4. Device Positioning and Removal (day 5)
5. Discharge/Final Visit (day 7-10)

Outcome Measures:

Primary Outcome Measures:

1. The difference in NIHSS between baseline and Day 7 vs. Historical Controls
2. % of patients with improvement in stroke symptoms (motor and/or sensory deficits) during stimulation

Additional Efficacy Outcome Measures:

1. Existence of physiologic surrogates of the Personal Stimulation Level
2. Improvement in stroke symptoms (motor and/or sensory deficits)

Safety Outcome Measures:

1. Comparative 7-day safety data between the ISS stimulation group of this study and of the ImpACT-24B study:

   1. Incidence of Serious Adverse Events
   2. Implantation Complications
   3. Stimulation-related Adverse Events
2. 7-day mortality
3. Neurological deterioration
4. Symptomatic intracranial hemorrhage (sICH)

Implantation Accuracy Outcome Measures:

1. % of procedures with positive indication of reaching the sphenopalatine fossa

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years and ≤ 80 years
2. Clinical diagnosis of anterior circulation stroke
3. Baseline NIHSS ≥ 1 and ≤ 6 or lacunar stroke of any severity
4. Motor and/or sensory deficits
5. Ability to initiate treatment within 24 hours from stroke onset
6. Signed informed consent from patient him/herself or legally authorized representative if applicable.

   Exclusion Criteria:
7. Neuro-imaging evidence of any intracranial hemorrhage or hemorrhagic transformation of brain infarct or other significant abnormality (e.g. tumor, abscess, suspect for subarachnoid hemorrhage).
8. Massive stroke, defined as acute parenchymal lesion with effacement of cerebral sulci in over 2/3 of the MCA territory.
9. Clinical signs and symptoms or evidence for a relevant lesion by neuro-imaging of an acute ischemic stroke in the posterior circulation (Vertebral, Basilar and/or Posterior Cerebral Artery territories), including but not limited to brain-stem findings and/or cerebellar findings and/or isolated homonymous hemianopia or cortical blindness.
10. NIHSS level of consciousness score ≥ 2.
11. Inability to communicate fluently and express symptoms
12. Previous motor and/or sensory deficits that will eliminate the ability to identify the response to SPG stimulation
13. Patients with bleeding propensity and/or one of the following: INR > 1.8, prolonged activated partial thromboplastin time (aPTT) ≥ 45 sec., platelets count < 75×109/L.
14. Known cerebral arteriovenous malformation, cerebral aneurysm.
15. Seizure at onset.
16. Blood glucose concentration < 60 mg/dL.
17. Clinical suspicion of septic embolus.
18. Uncontrolled hypertension (systolic >185 mmHg and/or diastolic >110 mmHg), demonstrated on each of three repeated measurements taken within one hour regardless of whether or not the patient is taking antihypertensive medications.
19. Serious systemic infection.
20. Women known to be pregnant or having a positive or indeterminate pregnancy test.
21. Patients with other implanted neural stimulator/ electronic devices (pacemakers).
22. History of SPG ablation ipsilateral to the stroke side.
23. Any condition in the oral cavity that prevents implantation of the INS, such as patient is intubated, orthodontics or non-hygienic condition.
24. Life expectancy < 1 year from causes other than stroke.
25. Participating in any other therapeutic investigational trial within the last 30 days.
26. Known sensitivity to any medications to be used during study.
27. Subjects who have a clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation. Conditions may include: cardiovascular, vascular, pulmonary, hepatic, renal or neurological (other than acute ischemic stroke), or neoplastic diseases, as determined by medical history, physical examination, laboratory tests, or ECG.
28. Subjects who, in the judgment of the investigator, are likely to be non- compliant or uncooperative during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
NIHSS Assessment | Day 7
  The difference in NIHSS between baseline and Day 7 vs. Historical Controls (the historical controls are patients in the control arm in the NINDS trial)
% of patients with improvement in stroke symptoms during stimulation | Day 2-5
  Assessment of improvement in stroke symptoms (motor and/or sensory deficits) before and during stimulation at the Personal Stimulation Level, using a hand dynamometer (Baseline Hydraulic Hand Dynamometers, Fabrication Enterprises Inc, White Plains NY, USA).

OTHER OUTCOMES:
Increased blood flow in Common Carotid Doppler | Day 1-5
  Increased blood flow in Common Carotid Doppler (if available) during stimulation at the Personal Stimulation Level (physiologic surrogates).
Existence of unilateral lacrimation, nasal secretion, and/or facial redness | Day 1-5
  Unilateral lacrimation, nasal secretion, and/or facial redness (on the stimulation side) during stimulation at the Personal Stimulation Level (physiologic surrogates).
Improvement in stroke symptoms | Day 2-5
  Assessment of improvement in stroke symptoms (motor and/or sensory deficits) before and during stimulation at the Personal Stimulation Level, using a hand dynamometer (Baseline Hydraulic Hand Dynamometers, Fabrication Enterprises Inc, White Plains NY, USA). The investigator will measure the grasp force and pincer force before and during stimulation in the affected and non-affected sides.

CONTACTS AND LOCATIONS:
Locations (4):
- Georgia (4):
  - Kutaisi Referral Hospital, Kutaisi
  - Rustavi Central Hospital, Rustavi
  - First University Clinic, Tbilisi
  - Zugdidi Referral Hospital, Zugdidi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saver JL, Kharaishvili N, Janelidze T, Beridze M, Zarqua N, Solberg Y, Bornstein NM; IMPACT-24M Trial Investigators. Refined Sphenopalatine Ganglion Stimulator Placement and Intensity Setting to Augment Blood Flow and Neurologic Function. Stroke. 2019 Dec;50(12):3512-3518. doi: 10.1161/STROKEAHA.119.027177. Epub 2019 Nov 19. PMID 31739771